CLINICAL TRIAL: NCT04447378
Title: Safety of Fondaparinux as Postpartum Venous Thromboembolism Prophylaxis
Brief Title: Safety of Fondaparinux as Post Partum Thromboprophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Aida Hani Mohd Kalok, Lecturer & Clinical Specialist, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEP -2017-543
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Thromboembolism in the Puerperium
Keywords: pregnancy; thromboembolism; prophylaxis
MeSH Terms: conditions — Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fondaparinux (Experimental): Subcutaneous injection of fondaparinux 2.5 mg once daily would be given over 10 days for post partum thromboprophylaxis
  Interventions: Drug: Fondaparinux 2.5Mg/0.5Ml Inj Syr

INTERVENTIONS:
Drug: Fondaparinux 2.5Mg/0.5Ml Inj Syr — post natal thromboprophylaxis
  Other Names: N/A; single arm study

SUMMARY:
Venous thromboembolism (VTE) remains as one of leading causes of maternal morbidity and mortality, with postpartum period carries the greatest risk. Perinatal thromboprophylaxis is often administered based on risk-factor assessment. Low molecular weight heparin has a proven safety profile in obstetrics population, however its porcine derived content may lead to reduced uptake amongst certain religious groups. The investigators aimed to evaluate the safety of fondaparinux as an alternative postpartum thromboprophylaxis.

The investigators planned a prospective, single arm, open label study. Women who fulfilled the criteria for post natal thromboprophylaxis based on the 2015 RCOG guidelines were recruited. Each patient would receive subcutaneous injection of Fondaparinux, 2.5mg daily for 10 days. The investigators would conduct a telephone interview on day 10 post delivery and six week outpatient review in clinic.

DETAILED DESCRIPTION:
All women were taught the injection technique and counselled regarding the symptoms of bleeding and VTE, prior to discharge. All patients were also advised to wear compression stockings and ensure adequate hydration at home

The primary outcome measure was occurrence of pulmonary embolism or deep vein thrombosis suggestive by clinical symptoms and assessment. Secondary outcome measures were allergic reaction and bleeding tendency such as secondary post-partum haemorrhage, spinal site bleeding and wound haematoma. Allergic reaction and bleeding tendency in neonates were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian
* Age 18 and above
* Scores asintermediate risk on 2015 Royal College of Obstetricians & Gynaecologists (RCOG) VTE risk assessment

Exclusion Criteria:

1. Hypersensitivity to fondaparinux
2. Patients with bleeding disorders - haemophilia , thrombocytopenia, von Willebrand's disease.
3. Weight < 50 kg
4. Patients with primary postpartum haemorrhage
5. Patients who already on anti - coagulants
6. Medical co morbidities - Systemic lupus erythematosus, heart failure, nephrotic syndrome, type 1 diabetes mellitus with nephropathy, sickle cell disease, current intravenous drug user
7. Uncontrolled hypertension ( blood pressure > 200 mmHg systolic or > 120 mmHg diastolic )

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism (VTE) | Within six weeks of delivery
  VTE occurence of either deep vein thrombosis or pulmonary embolism

SECONDARY OUTCOMES:
Major Bleeding requiring hospitalisation | within six weeks of delivery
  Secondary post partum haemorrhage or spinal site bleeding
Minor bleeding | within six weeks of delivery
  Wound site bleeding, skin bruising
Allergic reaction | within 24 hours from last injection
  Any allergy symptoms following injection of fondaparinux
Neonatal bleeding tendency | within six weeks of delivery
  Any bruising of bleeding tendency in neonates

CONTACTS AND LOCATIONS:
Overall Officials: Nor Azlin Mohamed Ismail, MBCHB, MMED, Principal Investigator — Faculty of Medicine, National University of Malaysia
Locations (1):
- Department of Obstetrics & Gynaecology, Universiti Kebangsaan Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD is available upon request